CLINICAL TRIAL: NCT00330382
Title: Bowman Birk Inhibitor Concentrate and Oral Leukoplakia: A Randomized Phase IIb Trial
Brief Title: Bowman-Birk Inhibitor Concentrate in Preventing Cancer in Patients With Oral Leukoplakia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00888; 98-34; U01CA072294 (NIH)
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-02

CONDITIONS: Lip and Oral Cavity Cancer; Oral Leukoplakia; Oropharyngeal Cancer; Tongue Cancer
MeSH Terms: conditions — Mouth Neoplasms; Leukoplakia, Oral; Oropharyngeal Neoplasms; Tongue Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (Bowman-Birk inhibitor concentrate) (Experimental): Patients receive oral Bowman-Birk inhibitor concentrate twice daily for 6 months
  Interventions: Drug: Bowman-Birk inhibitor concentrate; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive oral placebo twice daily for 6 months
  Interventions: Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Bowman-Birk inhibitor concentrate — Given orally
  Other Names: BBIC
  Arms: Arm I (Bowman-Birk inhibitor concentrate)
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well Bowman-Birk inhibitor concentrate works in preventing cancer in patients with oral leukoplakia. Chemoprevention is the use of certain substances to keep cancer from forming, growing, or coming back. The use of Bowman-Birk inhibitor concentrate, a substance made from soy, may keep cancer from forming in patients with oral leukoplakia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if chemoprevention by the Bowman-Birk inhibitor concentrate (BBIC) can prevent cancer in patients with oral leukoplakia (OL).

II. Determine the clinical and histologic response rate of OL to BBIC.

SECONDARY OBJECTIVES:

I. Measure the effect of BBIC on intermediate marker endpoint levels. II. Correlate the clinical and histologic responses of OL with cellular levels of proteolytic activity, erb-B2 (neu), retinioc acid receptor β, bcl-2, and mutant p53 expression, and serum levels of neu.

III. Determine the individual and group side effects of BBIC.

OUTLINE: This is a multicenter, randomized, double-blind, placebo-controlled, study. Prior to randomization, all patients receive oral placebo for 4 weeks. Patients who show good compliance (> 75% packet count) are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral Bowman-Birk inhibitor concentrate twice daily for 6 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive oral placebo twice daily for 6 months in the absence of disease progression or unacceptable toxicity.

Patients complete questionnaires about diet, tobacco, and alcohol usage at baseline and at the completion of study treatment. Blood, urine, and biopsy tissue are collected at baseline and at the completion of study treatment. Oral mucosal cells are collected at baseline, during the run-in phase, at randomization, after completion of study treatment, and at 3 months after completion of study treatment. Samples are examined for protease activity, levels of bcl-2 and erbB-2, mutant p53 oncogene expression and epidermal growth factor receptor, and retinoic acid receptor-β expression.

After completion of study treatment, patients are followed at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and clinically confirmed oral leukoplakia and/or erythroplakia
* Bidimensionally measurable disease (≥ 100 mm^2 for total area of all lesions) after biopsy
* No presence of obvious head and neck aerodigestive tract cancer, carcinoma in situ, or previously treated head and neck cancer within the past 2 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reaction to soybeans, sorbitol, sucrose, artificial flavorings, aspartame, saccharin, or lidocaine
* At least 6 months since prior Bowman-Birk inhibitor concentrate
* At least 6 months since prior participation in another randomized clinical trail
* At least 3 months since prior systemic steroids or topical oral steroid preparations

  * Topical nasal steroid sprays or cutaneous preparations with minimal systemic absorption for nasal or dermatologic disorders allowed
* More than 6 months since prior beta carotene capsules
* At least 2 years since prior retinoid or other beta carotene therapy, including > 25,000 IU of vitamin A for any reason

  * Up to 2 multivitamins per day allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 1999-01; Primary Completion 2010-07 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Meyskens, Principal Investigator — University of California Medical Center At Irvine-Orange Campus
Locations (1):
- University of California Medical Center At Irvine-Orange Campus, Orange, California, United States

REFERENCES:
- [Background] Meyskens FL. Development of Bowman-Birk inhibitor for chemoprevention of oral head and neck cancer. Ann N Y Acad Sci. 2001 Dec;952:116-23. doi: 10.1111/j.1749-6632.2001.tb02732.x. PMID 11795430
- [Background] Meyskens FL Jr. Development of difluoromethyl-ornithine and Bowman-Birk inhibitor as chemopreventive agents by assessment of relevant biomarker modulation: some lessons learned. IARC Sci Publ. 2001;154:49-55. PMID 11220668
- [Result] Armstrong WB, Taylor TH, Kennedy AR, Melrose RJ, Messadi DV, Gu M, Le AD, Perloff M, Civantos F, Goodwin WJ, Wirth LJ, Kerr AR, Meyskens FL Jr. Bowman birk inhibitor concentrate and oral leukoplakia: a randomized phase IIb trial. Cancer Prev Res (Phila). 2013 May;6(5):410-8. doi: 10.1158/1940-6207.CAPR-13-0004. PMID 23639862
- [Result] Armstrong WB, Wan XS, Kennedy AR, Taylor TH, Meyskens FL Jr. Development of the Bowman-Birk inhibitor for oral cancer chemoprevention and analysis of Neu immunohistochemical staining intensity with Bowman-Birk inhibitor concentrate treatment. Laryngoscope. 2003 Oct;113(10):1687-702. doi: 10.1097/00005537-200310000-00007. PMID 14520092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 513 people were screened for participation across all 8 performance sites, of which 188 (37%) were ineligible and 325 were consented.
Pre-assignment Details: Of 325 consented, 157 (48%) completed the run-in period but 25 declined to continue, resulting in 132 randomized patients.
Period: Overall Study
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo)
Started | 67 | 65
Completed | 43 | 48
Not Completed | 24 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo) | Total
Number analyzed (Participants) | 67 | 65 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.25 (13.63) | 60.64 (12.01) | 59.42 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Relative Percent Change in Total Lesion Area After 6 Months on Study
Description: Relative percent change in total lesion area was defined as 100 times (area posttreatment minus area pretreatment) all divided by pretreatment area.
Time Frame: 6 months
Population: The participants who have complete data are analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 46
percentage change | -20.6 (52.4) | -17.1 (66.4)

2. Secondary Outcome: The Difference in Rated Degree of Malignancy Between Randomization and 6-month Specimen
Description: The reviewer was blinded to study-arm assignment (drug or placebo), but not to time point of specimen. For each specimen, the reviewer marked a continuum to indicate degree of tissue abnormality. The continuum was 140 mm long, and anchored by the word 'Normal' on the left and 'Malignant' on the right. The distance from the left edge of the continuum to the reviewer's mark, in mm, was determined. For analyses, a score was formed by subtracting the pretreatment value from the 6-month value. Thus, a retreat from 'Malignancy' over time produces a negative score, a score of zero denotes no change, and a positive score denotes a worsening situation. Positive values indicate histologic worsening, whereas negative scores denote improvement over the 6-month study period.
Time Frame: Baselie to 6 months
Population: The participants who have complete data are analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo)
Number analyzed (Participants) | 41 | 47
score | 1.2 (23.7) | 3.6 (15.4)

3. Primary Outcome: Number of Participants by Category of Clinical Response at 6 Months
Description: Category of clinical response was based on the magnitude of relative percent change in total lesion area. A complete response (CR) was declared if the relative percent change in total lesion area was minus 100 percent. A partial response (PR) was a relative percent decrease in total lesion area of 50% or more, without being a CR. Disease progression was a relative percent increase in total lesion area of at least 50%. Remaining cases were declared to be stable disease.
Time Frame: 6 months
Population: The participants who have complete data are analyzed in this outcome measure.
Measure: Number; unit: participants
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 46
participants
  Complete response (CR) | 2 | 2
  Partial response (PR) | 10 | 12
  Stable disease | 27 | 26
  Disease progression | 4 | 6

4. Secondary Outcome: Clinical Impression From Photographs
Description: A secondary clinical response measure was bsaed on blinded, comparative judgments of pairs of photographs of the same lesion at baseline and 6 months on study. Picture pairs were assigned to album page, one pair per page, at random. Five physicians experienced with evaluation of oral mucosal tissue abnormalities, but blinded to study arm and time point, independently compared the pictures in each pair using a 7-point scale. The scale ranged from, "top photo shows a complete response relative to the bottom photo," through, "the same degree of disease is shown by top photo and bottom photo," to "bottom photo shows a complete response relative to the top photo." Raw scores were transformed to account for relative position of the earlier and later photo, and averaged across the 5 reviewers. Final scores ranged from one, denoting a CR at 6 months, to 4, which indicated no change, through 7, which indicated that the 6-month photo depicted a much worse situation than the pretreatment photo.
Time Frame: Baseline to 6 months
Population: The participants who have complete data are analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo)
Number analyzed (Participants) | 45 | 46
score | 4.0 (1.0) | 3.6 (0.9)

5. Secondary Outcome: Relative Percent Change in Buccal-Cell Neu Protein (ng/mg)
Description: 100% x (Posttreatment value - pretreatment value)/(pretreatment value)
Time Frame: Baseline to 6 months
Population: The participants who have complete data are analyzed in this outcome measure.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 24
percentage change | -10.1 [-52.3 to 24.6] | -4.2 [-33.6 to 36.7]

6. Secondary Outcome: Relative Percent Change in Serum Neu Protein (ng/ml)
Description: 100% x (Posttreatment value - pretreatment value)/(pretreatment value)
Time Frame: Baseline to 6 months
Population: The participants who have complete data are analyzed in this outcome measure.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 22
percentage change | -3.9 [-13.5 to 8.1] | -8.1 [-15.3 to 6.6]

7. Secondary Outcome: Relative Percent Change in Protease Activity (Delta RFU/Min/µg)
Description: 100% x (Posttreatment value - pretreatment value)/(pretreatment value)
Time Frame: Baseline to 6 months
Population: The participants who have complete data are analyzed in this outcome measure.
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 24
percentage change | 15.7 [-23.8 to 74.9] | 17.2 [-10.3 to 30.9]

8. Secondary Outcome: Number of Participants Report at Least 1 Adverse Event During the Study
Description: The onset of adverse event is between the randomizaiton date and off-study date
Time Frame: Randomized date to Off-study date, up to 21 months
Measure: Number; unit: participants
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo)
Number analyzed (Participants) | 67 | 65
participants
  Yes: report at least 1 AE | 33 | 25
  No: no AE reported | 34 | 40

9. Secondary Outcome: Combined Percentage Change From Baseline in Proteolytic Activity, Buccal-cell Erb-B2 (Neu) and Serum Levels of Neu at 6 Months
Time Frame: Baseline to 6 months
Population: The participants whose data are available and complete are included in the analysis.
Measure: Median (95% Confidence Interval); unit: percentage change
Groups:
- Combined Bowman-Birk Inhibitor Concentrate and Placebo Groups: Patients receive oral Bowman-Birk inhibitor concentrate or Placebo twice daily for 6 months
  Bowman-Birk inhibitor concentrate: Given orally Placebo: Given orally laboratory biomarker analysis: Correlative studies
Arm/Group | Combined Bowman-Birk Inhibitor Concentrate and Placebo Groups
Number analyzed (Participants) | 45
percentage change
  Buccal-Cell New | -8.9 [-24.5 to 18.5]
  Protease Activity | 16.2 [-10.0 to 27.0]
  Serum Neu (n=41) | -4.1 [-11.3 to 0.7]
Statistical Analysis 1: Comparison: Combined Bowman-Birk Inhibitor Concentrate and Placebo Groups; Correlation of percent change in buccal-cell Neu with relative percent change in total lesion area; Test type: Superiority or Other; p > 0.45, Spearman Rank Correlation; Correlation Coefficient = 0.11
Statistical Analysis 2: Comparison: Combined Bowman-Birk Inhibitor Concentrate and Placebo Groups; Correlation of percent change in protease activity with relative percent change in total lesion area; Test type: Superiority or Other; p > 0.88, Spearman Rank Correlation; Correlation Coefficient = 0.92
Statistical Analysis 3: Comparison: Combined Bowman-Birk Inhibitor Concentrate and Placebo Groups; Correlation of percent change in serum Neu with relative percent change in total lesion area; Test type: Superiority or Other; p > 0.66, Spearman Rank Correlation; Correlation Coefficient = 0.07

ADVERSE EVENTS:
Time Frame: The adverse-event reports were dated on or after randomization, up to 21 months.
Description: The number of adverse-event reports from the 132 randomized subjects dated on or after randomization was 138.
Arm/Group | Arm I (Bowman-Birk Inhibitor Concentrate) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 5/67 | 0/65
Other Adverse Events (participants affected / at risk) | 30/67 | 25/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Bowman-Birk Inhibitor Concentrate) (N=67) | Arm II (Placebo) (N=65)
ADMISSION FOR ORAL SURGERY ON FLOOR MOUTH (Surgical and medical procedures) | 1 (1) | 0 (0)
C/O "LUMP" TO RT. LOWER GUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLD (General disorders) | 1 (1) | 0 (0)
EPIGASTRIC PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
FINGER INFECTION - LEFT RING (Infections and infestations) | 1 (1) | 0 (0)
HEART PROBLEMS (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Bowman-Birk Inhibitor Concentrate) (N=67) | Arm II (Placebo) (N=65)
6 CROWNS (Surgical and medical procedures) | 1 (1) | 0 (0)
ABD PN AND BLOATING (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BAD BREATH (Gastrointestinal disorders) | 1 (1) | 0 (0)
BAD CANKER LOWER LIP (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BAD COLD (General disorders) | 0 (0) | 1 (1)
BLEEDING HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLOATED (Gastrointestinal disorders) | 1 (1) | 0 (0)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHITIS/FLU (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CAD (Cardiac disorders) | 1 (1) | 0 (0)
CANKER SORES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CARDIAC STENT (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOVASCULAR OTHER - GENERAL (Cardiac disorders) | 1 (2) | 0 (0)
CELLULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CHEST PAIN (Cardiac disorders) | 0 (0) | 2 (2)
CHIP FX ON RIGHT BIG TOE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COLD (General disorders) | 3 (3) | 1 (1)
COLD SORES (Infections and infestations) | 1 (1) | 0 (0)
COMPLAINED OF TASTE (Nervous system disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
CUT HAND WHILE PLAYING SOCCER AND NEEDED STITCHES (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DECREASED SEXUAL APPETITE (Psychiatric disorders) | 0 (0) | 1 (1)
DENTAL IMPLANTS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 3 (4) | 1 (1)
DIDN'T LIKE TASTE AFTER RUN IN AND THEN RANDOMIZED, STATED THAT HE "DIDN'T FEEL IT WAS WORKING". (Nervous system disorders) | 0 (0) | 1 (1)
DRY LIPS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
EAR INFECTION/IRREGULAR BUMP (Ear and labyrinth disorders) | 1 (1) | 0 (0)
EPIGASTRIC PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
EPIGASTRIC PAIN AND NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
FALL, COMPRESSION OF T11-L1 VERTEBRAL BODY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FISSURE FX (Gastrointestinal disorders) | 1 (1) | 0 (0)
FLU X 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
FLU X 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
FLU X 6 D (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
FLU/COLD (General disorders) | 0 (0) | 1 (1)
FNA AND BIOPSY OF MASS INTRAMUSCULAR LIPOMA (Surgical and medical procedures) | 1 (1) | 0 (0)
GAS-BUT THIS HAS DISAPPEARED AFTER BEING ON POWDER FOR ONE WEEK. (Gastrointestinal disorders) | 0 (0) | 1 (1)
GUM BLEEDING (Gastrointestinal disorders) | 0 (0) | 1 (2)
GUM EROSION (SONIC TOOTHBRUSH) (Gastrointestinal disorders) | 0 (0) | 1 (1)
GUMS FEEL SORE/TENDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
HANDS NUMB (Nervous system disorders) | 0 (0) | 1 (1)
HEAD COLD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHES (Nervous system disorders) | 1 (1) | 0 (0)
HIVES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HOSPITALIZAED RIGHT KNEE REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (1)
INCREASED HAIR LOSS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
INCREASED SENSITIVITY WITH SPICY FOOD, IE FROM MED TO MILD SALSA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INCREASED TONGUE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ITCHY FOREARM, POSSIBLE BUG BITE REACTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
KIDNEY STONES (Renal and urinary disorders) | 1 (2) | 0 (0)
LOOSE STOOLS (Gastrointestinal disorders) | 0 (0) | 1 (1)
LOWER LEFT JAW LESION FEELS ODD/STRETCHY (Psychiatric disorders) | 0 (0) | 1 (1)
LT. FOOT RUPTURED TENDON (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LT. FOOT THROMBUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LT. FOOT THROMBUS CONTINUES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
MASS 2-3 CM ON CT OF ABDOMEN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MOUTH SORES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
NAUSEA/ABD CRAMPING (Gastrointestinal disorders) | 0 (0) | 1 (1)
NEW SPOTS IN THROAT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ORAL SORENESS (General disorders) | 2 (3) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
POISON OAK (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PT FELL. LEFT EYEBROW AREA BRUISED (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
REDNESS OUTER ASPECT LIPS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ROOF OF MOUTH MORE SENSITIVE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RT HAND LITTLE FINGER BROKEN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SCIATIC LEG PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SCIATICA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SHINGLES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SINUS INFECTION, TOOK ZITHROMAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SOFT STOOL (Gastrointestinal disorders) | 2 (2) | 0 (0)
SORE - TONGUE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SORE MOUTH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SORE MOUTH - CORNERS AND GUMS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
SORE TONGUE BOTH SIDES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
STOMACH ACHE (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMACH DISTRESS WITH SPICY FOODS (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMACH FLU (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMACH PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
SURGERY ON FINGER (Surgical and medical procedures) | 0 (0) | 1 (1)
TASTED LIKE YEAST (Nervous system disorders) | 0 (0) | 1 (1)
TASTES BAD (Nervous system disorders) | 1 (1) | 0 (0)
THINNING HAIR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
THROAT DRY AND CHAULKY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
TIRED AND DIDN'T FEEL LIKE TAKING (Psychiatric disorders) | 1 (1) | 0 (0)
TIRED. IN RETROSPECT FELT TIRED DUE TO WORK. (General disorders) | 1 (1) | 0 (0)
TONGUE NUMBNESS COMES AND GOES (Nervous system disorders) | 1 (1) | 0 (0)
TONGUE NUMBNESS, TINGLING AND DRY MOUTH (Nervous system disorders) | 1 (1) | 0 (0)
TOOTH EXTRACTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTH INFECTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTH PULLED/EAR PAIN/ TOOTH DECAY (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOUNGE PAIN CONTINUES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TOUNGE SORENESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ULCERATION (SMALL) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ULCERATION X3 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
UNDERGOING ROOT CANAL (Surgical and medical procedures) | 1 (1) | 0 (0)
UPPER RESPIRATORY INFECTION AND SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
UPSET STOMACH (Gastrointestinal disorders) | 1 (1) | 1 (1)
UPSET STOMACH AND GAS (Gastrointestinal disorders) | 1 (1) | 0 (0)
URINARY FREQUENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
VOMITING - 2X THEN STOPPED (Gastrointestinal disorders) | 1 (1) | 0 (0)
WEIGHT LOSS 10LB DUE TO PAIN (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
YEAST INFECTION (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less